CLINICAL TRIAL: NCT01671865
Title: Magnetic Resonance Imaging and Spectroscopy Biomarkers for Facioscapulohumeral Muscular Dystrophy
Status: Active, not recruiting | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00065256
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
Keywords: FSHD; magnetic resonance imaging; magnetic resonance spectroscopy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research study is to identify and study changes in muscle in people with facioscapulohumeral muscular dystrophy using magnetic resonance imaging and spectroscopy.

DETAILED DESCRIPTION:
This research study is being done to study changes in muscle imaging over time in people with facioscapulohumeral muscular dystrophy (FSHD). Whole-body magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) will be used to evaluate skeletal muscle in study participants. This research is being done to assess how changes in muscle imaging correspond to muscle strength and function. Qualified participants will be asked to complete 5 study visits over 21 months. Each visit will include muscle strength and function testing in addition to the MRI/MRS scan. The investigators plan to use MRI and MRS in developing outcome measures that can be used in future clinical trials for FSHD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent for study participation (a parent or guardian will be asked to provide informed consent for participants younger than 18 years old)
* Confirmed diagnosis of FSHD through genetic testing (participants will be asked to provide copies of genetic testing results)

Exclusion Criteria:

* Any contraindication to MRI scanning
* Inability to complete a physical examination, including strength measurements

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include people with facioscapulohumeral muscular dystrophy confirmed through genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2012-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Intramuscular fat infiltration on MRI | Baseline, 3 months, 9 months, 15 months, and 21 months
  Intramuscular fat infiltration on MRI

SECONDARY OUTCOMES:
Intramuscular edema on MRI | Baseline, 3 months, 9 months, 15 months, and 21 months
  Intramuscular edema on MRI
Muscle strength testing | Baseline, 3 months, 9 months, 15 months, and 21 months
  Muscle strength testing
Timed function testing | Baseline, 3 months, 9 months, 15 months, and 21 months
  Timed function testing

CONTACTS AND LOCATIONS:
Overall Officials: Doris G Leung, MD, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Doris Leung, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung DG. Magnetic resonance imaging patterns of muscle involvement in genetic muscle diseases: a systematic review. J Neurol. 2017 Jul;264(7):1320-1333. doi: 10.1007/s00415-016-8350-6. Epub 2016 Nov 25. PMID 27888415
- [Background] Leung DG, Carrino JA, Wagner KR, Jacobs MA. Whole-body magnetic resonance imaging evaluation of facioscapulohumeral muscular dystrophy. Muscle Nerve. 2015 Oct;52(4):512-20. doi: 10.1002/mus.24569. Epub 2015 Mar 31. PMID 25641525
- [Background] Leung DG, Wang X, Barker PB, Carrino JA, Wagner KR. Multivoxel proton magnetic resonance spectroscopy in facioscapulohumeral muscular dystrophy. Muscle Nerve. 2018 Jun;57(6):958-963. doi: 10.1002/mus.26048. Epub 2018 Feb 14. PMID 29266323
- See also: Kennedy Krieger Institute Center for Genetic Muscle Disorders — https://www.kennedykrieger.org/patient-care/patient-care-centers/center-genetic-muscle-disorders